CLINICAL TRIAL: NCT06758284
Title: Effect of Laughter Yoga on Surgical Fear and Anxiety in Patients Applied Before Ureteroscopy: a Randomized Controlled Trial
Brief Title: Effect of Laughter Yoga on Surgical Fear and Anxiety in Patients Applied Before Ureteroscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Hatice Merve Alptekin, Research Assistant, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024/11/16
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Ureteroscopy; Kidney Stones
MeSH Terms: conditions — Kidney Calculi | interventions — Laughter Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laughter Yoga Group (Experimental): 1. 40 minutes before the procedure, the patients' surgical fear is evaluated.
  2. 40 minutes before the procedure, the patients' state anxiety is evaluated.
  3. A single session of laughter yoga is performed. (30 minutes)
  4. After laughter yoga, the patients' surgical fear is re-evaluated.
  5. After laughter yoga, the patients' state anxiety is re-evaluated.
  Interventions: Other: Laughter Yoga
- Control Group (No Intervention): 1. 40 minutes before the procedure, the patients' surgical fear is evaluated.
  2. 40 minutes before the procedure, the patients' situational anxiety is evaluated.
  1. 5 minutes before the procedure, the patients' surgical fear is evaluated. 2. 5 minutes before the procedure, the patients' situational anxiety is evaluated.

INTERVENTIONS:
Other: Laughter Yoga — The first component of the intervention is laughter therapy, which is a combination of warm-up exercises, deep breathing exercises, childlike playfulness and laughter exercises. Participants will do laughter therapy via WhatsApp video call. Laughter yoga will be a single session and will last approximately 30 minutes.
  Arms: Laughter Yoga Group

SUMMARY:
Surgical fear is a situation where a person experiences excessive fear of surgical procedures. This fear can negatively affect the person's normal life and is usually more intense in the pre-operative period. The causes of surgical fear include factors such as previous negative surgical experiences, lack of sufficient information, post-operative pain and complications. In addition, factors such as age, gender, and level of education can also affect fear. This fear can lead to physical and psychological problems along with stress; symptoms such as increased heart rate, dizziness, and muscle tension can be seen. Methods such as cognitive-behavioral therapy, meditation, and hypnosis can be used in the treatment of surgical fear. In addition, anxiety can also arise from thinking about the surgical procedure, post-operative complications, fear of anesthesia, or pain. High-risk surgeries and past negative experiences can increase anxiety. High anxiety before surgery can lead to psychological and physical problems. Nurses should offer anxiety-reducing techniques (breathing exercises, relaxation) by taking into account the needs of patients. In addition, having relatives with the patient can help relieve anxiety. Laughter yoga is considered an effective complementary therapy to reduce surgical fear and anxiety. Developed in India in 1995, this method involves simulating laughter with yoga breathing techniques. Laughter yoga relaxes muscles, increases pain threshold, and improves overall psychological well-being. This study aims to evaluate the effects of laughter yoga on patients undergoing ureteroscopy.

ELIGIBILITY:
Inclusion Criteria:

It will be applied to patients who agree to participate in the study, are scheduled to undergo ureteroscopy in a urological surgery clinic, have no hearing or vision problems, are over the age of 18, understand and speak Turkish, are literate, and can communicate.

Exclusion Criteria:

Patients with mental retardation and any psychiatric disorder, alcohol or drug addiction, hypertension or heart disease, hernia, glaucoma will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Surgical Fear | 40 minutes before the ureteroscopy procedure, 5 minutes before the ureteroscopy procedure
  The "Surgical Fear Questionnaire" will be used to measure patients' fear of surgery. The scale is an 11-point Likert-type scale consisting of 8 items, each item scored between 0 (not afraid at all) and 10 (very afraid). The scale has two sub-dimensions, each consisting of four items; items 1-4 measure fear of short-term outcomes of surgery, while items 5-8 measure fear of long-term outcomes of surgery. The sub-dimension scale score is obtained by summing the scores of each of the short-term and long-term sub-dimensions of the Surgical Fear Scale, and the total score of the scale is calculated by summing these scores. The sub-dimensions of the scale are scored between 0-40, and the total score is scored between 0-80. As the score increases, the patient's fear also increases.

SECONDARY OUTCOMES:
Anxiety | 40 minutes before ureteroscopy, 5 minutes before ureteroscopy
  Spielberg State-Trait Anxiety Inventory The scale consists of two separate dimensions: state anxiety (STAI-I) and trait anxiety (STAI-II), and these dimensions aim to measure individuals' anxiety in different contexts. The state anxiety section will be used in this study. The 20 items of the scale measure state anxiety. The scale items are in a 4-point Likert type. Responses range from "Never" (1) to "Very often" (4). The state anxiety scale contains 10 reverse (1, 2, 5, 8, 11, 15, 16, 19, 20) and 10 direct statements. The scale is scored between 20-80 and the anxiety level increases as the score increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsun Gazi State Hospital, Samsun, Samsun, Turkey (Türkiye)